## Phone Coaching for Weight Loss Maintenance Statistical Analysis Plan NCT04293055

Last Updated: 6/6/2024

**Statistical Plan.** Descriptive statistics will be used to compare the coaching and the control groups. Only individuals who regained 1.5% of their weight and triggered randomization will be included in the subsequent analysis, given the focus of the study is to compare conditions for individuals who experience weight regain. For the primary outcome (e.g., change in percent weight from baseline to 12 months), linear regressions predicting change in percent weight from baseline to 12 months controlling for baseline weight will be utilized. For the secondary outcome (e.g., percent weight change during the 40-day coaching window), linear regressions predicting change in percent weight from trigger day to 40 days post-trigger day controlling for trigger-day weight. Multiple imputation will be used to handle missing data.